CLINICAL TRIAL: NCT05880771
Title: Immediate Implant Placement: a Clinical and Radiographic Study on Hard and Soft Tissues Retraction at One Year.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Christian Makary, Professor, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XFMD203
Record Dates: First submitted 2023-05-14; First posted 2023-05-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-07

CONDITIONS: Immediate Implant Placement; Guided Surgery; Immediate Tamporization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate implant placement with buccal gap grafted with Allograft (Experimental): Following tooth extraction immediate implant will be placed in the palatal bone and the buccal gap between the implant and the buccal bone will be grafted with Allograft
  Interventions: Other: Immediate Implant Placement
- Immediate implant placement with buccal gap grafted with Xenograft (Experimental): Following tooth extraction immediate implant will be placed in the palatal bone and the buccal gap between the implant and the buccal bone will be grafted with Xenograft
  Interventions: Other: Immediate Implant Placement

INTERVENTIONS:
Other: Immediate Implant Placement — Tooth extraction followed by immediate implant placement. One group will have Allograft graft in the buccal gap, the other will have Xenograft graft.

SUMMARY:
This project consists of placing dental implants at extraction sites. Bone drilling and implant placement are performed using the flapless method with the use of a surgical guide allowing guided surgery. After implant placement, temporary teeth are immediately made and placed on the implants to guide the gingival contour.

Bone and soft tissue retraction at the implanted sites are measured radiographically and digitally using surface scan superimposition over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Absence of systemic or osseous disease that may impair peri-implant healing
* Age ≥ 21 years
* Acceptable oral hygiene
* Presence of both adjacent teeth
* Absence of acute infection in the treated area
* Absence of periodontal pockets > 3mm at the concerned site
* Absence of pre-operative defect at the buccal bone wall (dehiscence or fenestration)
* Per-operative integrity of the osseous and gingival structures (during tooth extraction)
* Light or non-smoker (<10 cigarettes per day)

Exclusion Criteria:

* Myocardial infarction within the past 6 months.
* Poorly controlled diabetes (HBA1c > 7.5%).
* Coagulation disorders.
* Radiotherapy to the head/neck area within the past two years.
* Present or past treatment with intravenous bisphosphonates.
* Immunocompromised patients.
* Psychological or psychiatric problems.
* Alcohol or drug abuse.
* Poor oral hygiene and motivation (full mouth plaque score > 30% and/or full mouth bleeding score > 20%).
* Uncontrolled periodontal disease.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Hard tissue change by superimposing CBCT scans between 0 and 12 months using 3d slicer software | 12 months
  Buccal bone profil retraction after immediate implant placement using 2 different bone substitutes by comparing CBCT Dicom files at 0 and 12 months using 3d slicer software
Soft tissue change by superimposing surface intraoral scans between 0 and 12 months using 3d slicer software | 12 months
  Soft Tissue profil retraction after immediate implant placement using 2 different bone substitutes by superimposing STL files between 0 and 12 monts using 3d slicer software

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided